CLINICAL TRIAL: NCT05350631
Title: Efficacy Study on Quality of Life Criteria of a Digital Application on Any Cellphone (OnKO-Tips&Tricks) Allowing Daily Follow-ups, Implementation of an ETP Program and a Direct Link With the Nurse Coordinator of Units Specifically Dealing With Adolescents and Young Adults Diagnosed With Cancer
Brief Title: Efficacy Study on Quality of Life Criteria of a Digital Application on Any Cellphone (OnKO-Tips&Tricks) for Adolescents and Young Adults Diagnosed With Cancer
Acronym: OnKO T&T 2 0
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 8360
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Adolescents population; Young adults population
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): only follow-ups consultations, phone contact and TVE workshop with the AJA mobile team centralized by the IDEC
- Experimental (Experimental): using a digital tool in addition to follow-ups by consultations, phone contact and PTE workshop with the AJA mobile team centralized by the IDEC
  Interventions: Other: OnKO-Tips&Tricks digital phone application

INTERVENTIONS:
Other: OnKO-Tips&Tricks digital phone application — Using daily OnKO-Tips&Tricks digital phone application
  Arms: Experimental

SUMMARY:
Approximately 2,200 cancers per year in France are diagnosed within the adolescents and young adults population (15-25 years old, AYA). The cancer plans and the INCA recommend support during and after cancer treatment, taking into account both medical and psycho-social specificities related to age (support care, school learning/training and professional integration, fertility preservation, therapeutic education, addictology, sexology...). In this context, AJA teams have been developed in which the Nurse Coordinators (IDEC) play a fundamental role. These Nurse Coordinators are available to young patients, their families and the professionals who accompany follow them in their therapeutic journey. Their main missions are to assess the specific needs of these young people and their loved ones, to inform, orient and participate in the coordination of their care by providing psychosocial and paramedical solutions to these young patients. The circular of 30/05/2016 on the coordinated regional organization of care for AJAs supports the development of connected health tools for AJAs. This population is adept to new technologies, social networks allowing them to continue to be informed and remain integrated to the outside world while helping them prepare for life after cancer.

In this context, our team initiated the development of a digital application compatible for any cellphone OnKO-Tips&Tricks meeting these criteria of necessity with the company CAPCOD. We would want to move on to a validation stage by carrying out a national multicenter efficacy study in AJA mobile units by comparing two groups of patients: users/non-users of this digital tool on a main criterion of quality of life after using it for 6 months. As it should promote autonomy and integration into the care pathway as well as active participation in therapeutic education programs (TPE), these different items will be evaluated as secondary endpoints of our study

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 15 years and ≤ 25 years
* Diagnosed with solid or blood cancers less than 1 month old or patient with relapsed cancer more than 5 years after completion of initial treatment
* Follow-up at one of the participating study centers
* Informed and signed consent from the patient and, if the subject is a minor, from the holders of parental authority
* Inclusion in the study at the latest at the time of initiation of chemotherapy or radiotherapy
* Patient agrees to 12-month post-inclusion follow-up
* Patient agreeing to complete all study questionnaires
* Patient with a cellphone capable of downloading the app (developed for all types of cellphones)
* Affiliated to a social health insurance plan

Exclusion Criteria:

* Patient deprived of liberty by a judicial or administrative decision
* Patient with protected person status
* Patient who does not understand, speak or write French
* Patient unable to understand the follow-up protocol according to the investigating physician or the IDEC of the AJA unit
* Patient with a scheduled hospitalization of at least 5 weeks during study participation

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of the OnKO-Tips&Tricks digital phone application on the psychosocial dimension of patients' quality of life | 6 months of inclusion
  Assessed using a psychosocial health score obtained by the Pediatric Quality of Life Inventory™ Version 4.0 Generic Core Scales questionnaire.
  The PedsQL 4.0 Generic Core Scale contains 23 items that measures physical (eight items), emotional (five items), social (five items), and school (five items) functions. The Scale comprises parallel patient self-report and parent proxy-report formats. The items are reverse-scored and trans- formed to a 0-100 scale according to the instructions, and higher scores indicate a better HRQOL.

SECONDARY OUTCOMES:
Evaluate the efficacy of the OnKO-Tips&Tricks digital phone application on the psycho-social dimension of patients' quality of life | 3 months and 12 months of inclusion
  Assessed using a psychosocial health score obtained from the Pediatric Quality of Life Inventory™ Version 4.0 Generic Core Scales questionnaire.
  The PedsQL 4.0 Generic Core Scale contains 23 items that measures physical (eight items), emotional (five items), social (five items), and school (five items) functions. The Scale comprises parallel patient self-report and parent proxy-report formats. The items are reverse-scored and trans- formed to a 0-100 scale according to the instructions, and higher scores indicate a better HRQOL.
Evaluate the efficacy of the OnKO-Tips&Tricks digital phone application on patients' overall and physical quality of life | 3 months, 6 months and 12 months of inclusion
  Assessed using total Quality of Life and physical health subscore scores obtained from the Pediatric Quality of Life Inventory™ Version 4.0 Generic Core Scales questionnaire.
  The PedsQL 4.0 Generic Core Scale contains 23 items that measures physical (eight items), emotional (five items), social (five items), and school (five items) functions. The Scale comprises parallel patient self-report and parent proxy-report formats. The items are reverse-scored and trans- formed to a 0-100 scale according to the instructions, and higher scores indicate a better HRQOL.
Evaluate the impact on each patient's participation in a therapeutic education program (TPE) | through study completion, an average of 1 year and 6 months
  Rate of patients in the experimental and control groups who will participate in the proposed FTE program
Evaluate the efficacy of the OnKO-Tips&Tricks digital phone application throughout the patient's care pathway | 3 months, 6 months and 12 months of inclusion
  assessed by the number of consultations, medical and paramedical, the number of outpatient management, the number of unscheduled hospitalizations, the number of listed side effects, and the number of phone contacts (text, calls) and emails initiated by the patient towards the IDEC.
Assess patient satisfaction with the use of the OnKO-Tips&Tricks digital phone application using the MAUQ questionnaire | 6 and 12 months
  Evaluated using the mHealth app usability questionnaire (MAUQ questionnaire).
Evaluate the adherence to the application in the experimental group | Per week and per month through study completion, an average of 1 year and 6 months
  Evaluated by collecting the number of uses of each feature
Evaluate the efficacy of the OnKO-Tips&Tricks digital phone application on the quality of life of patients according to cancer pathology | 6 months of inclusion
  Comparative analysis of quality of life collection using the Pediatric Quality of Life Inventory™ Version 4.0 Generic Core Scales questionnaire taking into account the type of cancers: solid vs. blood cancer The PedsQL 4.0 Generic Core Scale contains 23 items that measures physical (eight items), emotional (five items), social (five items), and school (five items) functions. The Scale comprises parallel patient self-report and parent proxy-report formats. The items are reverse-scored and trans- formed to a 0-100 scale according to the instructions, and higher scores indicate a better HRQOL.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Institut d'Hématologie et d'Oncologie Pédiatrique, Lyon, France
  - Hôpital enfant-adolescent, Nantes, France
  - CHU de Nice Hôpital Archet 2, Nice, France
  - CHU Reims - Hôpital Maison Blanche, Reims, France
  - Hôpitaux Universitaires de Strasbourg, Strasbourg, France
  - Assistance Publique - Hôpitaux de Marseille, Marseille
  - CHU Rennes Hôpital Sud, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de Cancerologie Strasbourg Europe, Strasbourg
  - Institut Gustave Roussy, Villejuif